CLINICAL TRIAL: NCT00263250
Title: Watchful Waiting Versus Open Tension-free Repair of Inguinal Hernia in Asymptomatic or Minimally Symptomatic Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01HS009860 (AHRQ)
Record Dates: First submitted 2005-12-06; First posted 2005-12-08 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; asymptomatic; watchful waiting; tension-free hernia repair
MeSH Terms: conditions — Hernia, Inguinal | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: watchful waiting or tension-free hernia repair

SUMMARY:
This is a multicenter clinical trial to compare pain, physical function, and other outcomes in men with asymptomatic or minimally symptomatic inguinal hernias randomly assigned to watchful waiting without an operation, or a standard hernia repair with mesh. We studied the safety of delaying operation.

DETAILED DESCRIPTION:
CONTEXT Many men with an inguinal hernia have minimal symptoms. Whether deferring operation is safe and a good option for some patients has not been assessed.

OBJECTIVE To compare pain and the Physical Component Score (PCS) of the SF-36 at two years in men with minimally symptomatic inguinal hernias randomized to watchful waiting (WW) or a standard tension-free hernia repair (TFR).

DESIGN, SETTING, AND PATIENTS. Between January, 1999 and December, 2004 we conducted a multicenter trial of 720 men (364 WW, 356 TFR) who were followed for 2-4.5 years. Men were excluded with hernia pain interfering with activities; undetectable hernias; infection; American Society of Anesthesiologists Physical Status >3; recent difficulty in reducing the hernia.

INTERVENTIONS Men assigned to WW were followed at 6 months and annually and watched for hernia symptoms. Men assigned to operation received TFR, and were followed at 3 and 6 months, and annually.

ELIGIBILITY:
Inclusion Criteria: men 18 years of age and older with asymptomatic or minimally symptomatic inguinal hernias who give informed consent to be randomized.

-

Exclusion Criteria:Presence of pain limiting usual activities, difficulty in reducing hernia within last 6 weeks, undetectable hernias, local or systemic infection, ASA physical status >3, or participation in another clinical trial.

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724
Dates: Start 1999-02; Primary Completion 2004-12 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Pain limiting usual activities at two years.
Physical function (PCS) at two years.

SECONDARY OUTCOMES:
Complications
patient-reported outcomes of pain, functional status, activity levels, and satisfaction with care.
Cost effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Jonasson, M.D., Study Director — American College of Surgeons
Locations (1):
- American College of Surgeons, Chicago, Illinois, United States

REFERENCES:
- [Result] Fitzgibbons RJ Jr, Giobbie-Hurder A, Gibbs JO, Dunlop DD, Reda DJ, McCarthy M Jr, Neumayer LA, Barkun JS, Hoehn JL, Murphy JT, Sarosi GA Jr, Syme WC, Thompson JS, Wang J, Jonasson O. Watchful waiting vs repair of inguinal hernia in minimally symptomatic men: a randomized clinical trial. JAMA. 2006 Jan 18;295(3):285-92. doi: 10.1001/jama.295.3.285. PMID 16418463
- [Derived] Schroeder AD, Tubre DJ, Fitzgibbons RJ Jr. Watchful Waiting for Inguinal Hernia. Adv Surg. 2019 Sep;53:293-303. doi: 10.1016/j.yasu.2019.04.014. Epub 2019 May 15. No abstract available. PMID 31327453
- [Derived] Ramanan B, Maloley BJ, Fitzgibbons RJ Jr. Inguinal hernia: follow or repair? Adv Surg. 2014;48:1-11. doi: 10.1016/j.yasu.2014.05.017. PMID 25293603
- [Derived] Fitzgibbons RJ Jr, Ramanan B, Arya S, Turner SA, Li X, Gibbs JO, Reda DJ; Investigators of the Original Trial. Long-term results of a randomized controlled trial of a nonoperative strategy (watchful waiting) for men with minimally symptomatic inguinal hernias. Ann Surg. 2013 Sep;258(3):508-15. doi: 10.1097/SLA.0b013e3182a19725. PMID 24022443
- [Derived] Sarosi GA, Wei Y, Gibbs JO, Reda DJ, McCarthy M, Fitzgibbons RJ, Barkun JS. A clinician's guide to patient selection for watchful waiting management of inguinal hernia. Ann Surg. 2011 Mar;253(3):605-10. doi: 10.1097/SLA.0b013e31820b04e9. PMID 21239979
- See also: American College of Surgeons — http://www.facs.org